CLINICAL TRIAL: NCT07198659
Title: A Single-Arm Investigator-Initiated Tria (IIT) Evaluating the Safety and Preliminary Efficacy of Autologous Drug-Loaded Neutrophils (NeuMed) in Patients With Unresectable Pancreatic Cancer（NeuMed-uPC）
Brief Title: A Single-Arm Investigator-Initiated Tria (IIT) Evaluating the Safety and Preliminary Efficacy of Autologous Drug-Loaded Neutrophils (NeuMed) in Patients With Unresectable Pancreatic Cancer
Acronym: NeuMed-uPC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Air Force Medicial University (Other)
Responsible Party: Principal Investigator, Lin Wang, Professor, The First Affiliated Hospital of Air Force Medicial University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252120
Record Dates: First submitted 2025-08-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Unresectable Pancreatic Cancer
Keywords: Autologous Drug-Loaded Neutrophils (NeuMed); Unresectable Pancreatic Cancer; Monomethyl Auristatin E (MMAE)
MeSH Terms: interventions — monomethyl auristatin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monomethyl Auristatin E (MMAE) / autologous neutrophil biological agents (Experimental): Isolate the patients' autologous neutriphil cells, induce and culture them with Monomethyl Auristatin E (MMAE) in a GMP-compliant laboratory. Prior to the reinfusion of neutrophil biological agents into patients, stereotactic radiotherapy with a dose of 2-6 Gy is administered to pancreatic cancer lesions. The number of neutrophils that were reinfused was 2.0-8.0x10^8.
  Interventions: Combination Product: Monomethyl Auristatin E (MMAE) / autologous neutrophil biological agents

INTERVENTIONS:
Combination Product: Monomethyl Auristatin E (MMAE) / autologous neutrophil biological agents — Isolate the patients' autologous neutriphil cells, induce and culture them with Monomethyl Auristatin E (MMAE) in a GMP-compliant laboratory. Prior to the reinfusion of neutrophil biological agents into patients, stereotactic radiotherapy with a dose of 2-6 Gy is administered to pancreatic cancer lesions. The number of neutrophils that were reinfused was 2.0-8.0x10^8.

SUMMARY:
The goal of this clinical trial is to learn if Autologous Drug-Loaded Neutrophils (NeuMed) can treat patients with Unresectable Pancreatic Cancer. The drug carried by the Autologous Neutrophils is Monomethyl Auristatin E. The main questions it aims to answer are: First, to verify the safety of Autologous Drug-Loaded Neutrophils (NeuMed) in patients with Unresectable Pancreatic Cancer. Second, to assess the anti-tumor efficacy of Autologous Drug-Loaded Neutrophils (NeuMed) in patients with Unresectable Pancreatic Cancer.

DETAILED DESCRIPTION:
In this open, single-armed study, selected patients with Unresectable Pancreatic Cancer confirmed by Histopathology will be received Autologous Drug-Loaded Neutrophils (NeuMed)-based therapy. Neutrophils will be isolated using a blood cell separator and cultured in a GMP-compliant laboratory to prepare neutrophil biological agents, which will then be loaded with the anti-tumor peptide, Monomethyl Auristatin E (MMAE).

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* Obtain an informed consent form voluntarily signed by the patient themselves
* patients with Unresectable Pancreatic Cancer confirmed by Histopathology
* Patients who either: 1) have received standard first-line treatments, proven ineffective or causing intolerable adverse effects; or 2) have not received the standard first-line treatments and voluntarily opt for Autologous Drug-Loaded Neutrophils (NeuMed)-based therapy
* EOCG score ≤ 2 and expected survival time ≥ 3 months
* Liver, kidney and bone marrow functions are basically normal

Exclusion Criteria:

* Patients who required anti coagulant therapy
* Patients with active infectious diseases or a history of bone marrow or organ transplantation
* Patients with autoimmune diseases or autoinflammatory diseases
* Patients with a history of severe cardiovascular or cerebrovascular diseases or interstitial lung disease or non-infectious pneumonia
* Patients who have received live vaccines within 30 days prior to enrollment
* Patients with no response to bone marrow mobilization
* Other patients deemed unsuitable for enrollment by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-07-14 (Estimated); Study Completion 2027-07-14 (Estimated)

PRIMARY OUTCOMES:
To verify the safety of Autologous Drug-Loaded Neutrophils (NeuMed) in patients with Unresectable Pancreatic Cancer | 12 months
  Incidence rate of Adverse Events（For the grading of treatment-related adverse events, all cases were classified with reference to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)）.
  Developed by the National Cancer Institute (NCI), the Common Terminology Criteria for Adverse Events (CTCAE) is currently the most widely used adverse event (AE) grading system, applicable to oncology clinical trials. It classifies adverse events into 5 grades:Grade 1 (Mild): Asymptomatic or mild in severity, with no requirement for intervention;Grade 2 (Moderate): Requiring medical intervention and causing mild impairment of daily activities;Grade 3 (Severe): Resulting in significant functional impairment, necessitating hospitalization or substantial medical intervention, and rendering the patient unable to perform daily activities;Grade 4 (Life-threatening): Pose a threat to life and require urgent intervention;Grade 5 (Death): Directly caused by the adverse event.

SECONDARY OUTCOMES:
To assess the anti-tumor efficacy of Autologous Drug-Loaded Neutrophils (NeuMed) in patients with Unresectable Pancreatic Cancer | 12 months
  Objective Response Rate (ORR)；The ORR is determined by measuring the size of target and non-target tumor lesions in follow-up imaging data, in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST).
  The Response Evaluation Criteria in Solid Tumors (RECIST) classifies tumor response to treatment into distinct categories based on changes in the size of target lesions (and non-target lesions, as applicable) and the presence of new lesions, with the following specific grading framework:Complete Response (CR)；Partial Response (PR)；Stable Disease (SD)；Progressive Disease (PD). Imaging modalities for lesion measurement (e.g., contrast-enhanced CT, MRI) must be consistent throughout follow-up to ensure the reliability of SLD calculations, as mandated by the specific grading criteria in RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Wang, Doctor of Medicine(M.D.), Study Director — The First Affiliated Hospital of Air Force Military Medical University; Liang Jin, Doctor of Medicine(M.D.), Principal Investigator — The First Affiliated Hospital of Air Force Military Medical University; Yong Chen, Doctor of Medicine(M.D.), Principal Investigator — The First Affiliated Hospital of Air Force Military Medical University
Locations (1):
- The First Affiliated Hospital of the PLA Air Force Military Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No